CLINICAL TRIAL: NCT01918943
Title: Evaluation of Aspen Spinous Process Fixation System and PLIF Technique for the Treatment of Low Back Pain in the Presence of Lumbar Instability and Degenerative Disk Disease
Brief Title: Evaluation of Aspen Spinous Process Fixation System and PLIF Technique for the Treatment of Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: American British Cowdray Medical Center (Other)
Responsible Party: Principal Investigator, Galvan Ernesto Eduardo, MD, American British Cowdray Medical Center
Other Study IDs: ABC-Aspen-2013
Record Dates: First submitted 2013-08-06; First posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Low Back Pain; Spondylolisthesis; Spondylosis; Spinal Instability; Spinal Stenosis
Keywords: Spine; Aspen device; PLIF; Low back pain
MeSH Terms: conditions — Low Back Pain; Spondylolisthesis; Spondylosis; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PLIF and Aspen device patients: All patients will receive PLIF and Aspen device
  Interventions: Device: PLIF and Aspen (spinous process fixation device)

INTERVENTIONS:
Device: PLIF and Aspen (spinous process fixation device) — Circunferential fusion with PLIF and postero-lateral fusion with the Aspen device

SUMMARY:
Lumbar spinal fusion was introduced approximately 70 years ago and has evolved as a treatment option for symptomatic spinal instability, spinal stenosis, spondylolisthesis, and degenerative scoliosis.

Many techniques evolved since then, from wiring, rods, pedicle screws, and recently inter-spinous fixation devices like the Aspen. Along its evolutionary trail, various methods for achieving circumferential fusion have arisen. Distinct from staged anterior/posterior fusion techniques, two methods of achieving an interbody fusion from a posterior approach have emerged: posterior lumbar interbody fusion (PLIF) and transforaminal lumbar interbody fusion (TLIF). Recently, the lateral approach for interbody fusion (XLIF) has became a more common technique, requiring in some cases, complemental posterior fixation with pedicle screws, facet screws or interspinous fixation devices like the Aspen device.

In this study, we address the clinical and radiological outcome of a novel technique using standard PLIF interbody fusion and insertion of the Aspen device via posterior lumbar approach.

ELIGIBILITY:
Inclusion Criteria:

* Oswestry Disability Index score >30%
* Diagnosis of low back pain and/or radicular pain associated to spinal instability
* Diagnosis of low back pain and/or radicular pain associated to degenerative disc disease
* Elective single level surgery
* Signed informed consent form

Exclusion Criteria:

* Previous surgery with complete laminectomy, pars defect, etc
* Patients that during the surgery requires complete laminectomy at level of the surgery
* Structural lesion to facet joints
* Osteoporosis
* Systemic or local infection
* Pregnant or planning to become pregnant

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 40 years and older with clinical and radiological signs of low back pain and spinal instability or degenerative disc disease requiring single level decompression and fusion.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index Score Change | 12 months
  Change between Oswestry Disability Index between pre-operative and final 12 months socores

SECONDARY OUTCOMES:
Rolland Morris Score | 12 months
  Change in score in the Rolland Morris Score (RMS)
Visual Analogue Scale | 12 months
  Change in pain measured by the visual analogue scale
Bone fusion (arthrodesis) | 12 months
  Adequate bone fusion measured by computed tomography (CT) scan

OTHER OUTCOMES:
Operative parameters | At surgery
  Surgery time, blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Roberto De Leo Vargas, MD, Study Director — Centro Medico ABC; Maximino Tellez, MD, Study Chair — Centro Medico ABC; Rodrigo Navarro, MD, Study Chair — Centro Medico ABC
Locations (1):
- American British Cowdray Medical Center, Mexico City, Mexico DF, Mexico